CLINICAL TRIAL: NCT06696690
Title: The Safety and Efficacy of Median Nerve Electrical Stimulation for Improving Neurological Function Prognosis in Patients With Cardiac Arrest: A Multicenter, Prospective, Randomized Controlled Study
Brief Title: The Safety and Efficacy of Median Nerve Electrical Stimulation for Improving Neurological Function Prognosis in Patients With Cardiac Arrest
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tang Ziren (Other)
Responsible Party: Sponsor-Investigator, Tang Ziren, Professor, Capital Medical University
Organization: Capital Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2024-6-7-3
Record Dates: First submitted 2024-11-17; First posted 2024-11-20 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Median Nerve; Coma; Post Cardiac Arrest Brain Injury
MeSH Terms: conditions — Coma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MNS treatment group (Experimental): Bundle treatment after cardiac arrest. Meanwhile, use the NeuroTrac™ Multi-TENS transcutaneous electrical stimulator to provide an asymmetric biphasic pulse train with a frequency of 35 Hz, an amplitude of 20 mA and a pulse width of 300ms, which is on for 20 seconds and off for 50 seconds. The treatment lasts for 8 hours per day and the treatment course lasts for 14 days.
  Interventions: Device: MNS
- Sham stimulation treatment group (Placebo Comparator): Bundle treatment after cardiac arrest. The control group utilized the same stimulation device and was subjected to a safe yet ineffective stimulation protocol for sham stimulation. The treatment lasts for 8 hours per day and the treatment course lasts for 14 days.
  Interventions: Device: Sham stimulation

INTERVENTIONS:
Device: MNS — The MNS treatment group use the NeuroTrac™ Multi-TENS transcutaneous electrical stimulator to provide an asymmetric biphasic pulse train with a frequency of 35 Hz, an amplitude of 20 mA and a pulse width of 300 ms, which is on for 20 seconds and off for 50 seconds. The treatment lasts for 8 hours per day and the treatment course lasts for one week.
  Arms: MNS treatment group
Device: Sham stimulation — The sham stimulation treatment group utilized the same stimulation device and was subjected to a safe yet ineffective stimulation protocol for sham stimulation. The treatment lasts for 8 hours per day and the treatment course lasts for 14 days.
  Arms: Sham stimulation treatment group

SUMMARY:
Median nerve stimulation (MNS), a non-invasive brain stimulation technique, has been widely adopted in clinical arousal therapies and multiple clinical investigations have attested to the efficacy of this technique; nevertheless, evidence concerning the application of MNS in improving the neurological prognosis of patients with return of spontaneous circulation (ROSC) following cardiac arrest (CA) remains scarce. The current study endeavors to assess the safety and efficacy of MNS treatment in enhancing the neurological prognosis of CA patients after ROSC and it is designed as a multicenter, prospective, randomized controlled trial with an estimated sample size of 400 patients. Eligible patients will be randomly allocated in a 1:1 ratio to either receive MNS treatment or sham stimulation treatment for 8 hours per day for 14 consecutive days and the primary outcome measure is the proportion of patients in each group with a Cerebral Performance Category (CPC) score ranging from 1 to 2, 6 months after randomization, which will help to determine the effectiveness of MNS in providing neuroprotection for patients with ROSC after CA.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old.
2. Hemodynamics remains continuously stable for ≥ 7 days.
3. There is still a lack of purposeful movements after the return of spontaneous circulation following cardiopulmonary resuscitation.
4. Advanced life support is provided within 6 hours after the return of spontaneous circulation (ROSC).

Exclusion Criteria:

1. Patients with hemodynamic instability.
2. Pregnant patients.
3. Those who have abnormal anatomical structures on the median nerve conduction pathway and are unable to receive electrical stimulation.
4. Patients with a confirmed history of epilepsy before admission or during hospitalization.
5. Patients with severe arrhythmia or those who have pacemakers implanted.
6. Patients whose family members do not agree to their enrollment in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients with a CPC score of 1-2 | 180 days
  The primary outcome is the proportion of patients with a score of 1-2 at 180 days after randomization in each group. Favorable: 1 means full recovery or mild disability; 2 means moderate disability but independent in activities of daily living (ADLs). Unfavorable: 3 means severe disability-Dependent in ADLs; 4 means persistent vegetive state; 5 means Death.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Chao-Yang Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Starting 6 months after publication
Access Criteria: The de-identified survey data will be made available for research purposes by contacting the corresponding authors